CLINICAL TRIAL: NCT06116188
Title: Brain Insulin Resistance in Mild Cognitive Impairment
Acronym: COINS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 57 /1801/2022
Record Dates: First submitted 2023-10-17; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Positron Emission Tomography
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: None Retained — Plasma and urine samples for measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Mild cognitive impairment: 20 study volunteers with a diagnosis of MCI due to AD or early AD or episodic memory decline during the last 6 months from the local memory clinics and by contacting doctors who treat and diagnose memory disorders. Patients with Alzheimer´s dementia - i.e. cognitive impairment severe enough to cause problems in activities of daily living - will not be included in the study due to the study protocol which requires co-operation and the ability to lie still in the PET scanner for approximately 60 minutes.
  Interventions: Diagnostic Test: FDG-PET study
- Healthy controls: We will also recruit 20 cognitively unimpaired controls, matched for age and gender for the patients group.
  Inclusion criteria for the cognitively unimpaired group for the present study are:
  i) no subjective cognitive complaints ii) CERAD (consortium to establish a registry for Alzheimer´s Disease) test battery at screening visit: CERAD total score within the normal range iii) clinical dementia rating (CDR) = 0, based on an interview with the study volunteer´s spouse or close relative iv) age 55 to 80 years
  Interventions: Diagnostic Test: FDG-PET study

INTERVENTIONS:
Diagnostic Test: FDG-PET study — Hyperinsulinemic, euglycemic clamp technique will be used to promote tissue glucose uptake and measure insulin sensitivity. Two cannulas will be inserted, one in a radial or an antecubital vein for PET tracer injection and infusion of glucose and insulin, another in the opposite radial or antecubital vein for blood sampling. In the clamp study subjects are administered intravenous insulin at a steady rate of 40 mU/m2/min and normoglycemia is maintained using a variable rate infusion of 20% glucose based on plasma glucose measurements, which are performed every 5min from arterialized venous blood. We will also collect samples to determine plasma insulin, serum free fatty acid and metabolic biomarkers during the study.
  The clamp will be performed together with [18F]-FDG-PET/CT.

SUMMARY:
Alzheimer´s disease (AD) is the most common cause of dementia. The most important risk factor for AD is old age; modifiable risk factors for AD include metabolic risk factors, i.e. diabetes, and obesity. Insulin resistance seems to be associated with AD pathology and cognitive decline. Previous studies suggest that AD and mild cognitive impairment (MCI) due to AD, a stage between normal cognition and AD dementia, would be associated with central nervous system (CNS) insulin resistance.

Insulin resistance can be measured using a sophisticated hyperinsulinemic-euglycemic clamp technique. Insulin-stimulated glucose uptake of muscles and adipose tissue is known to be reduced in an insulin resistant subject compared to healthy insulin sensitive subjects. Central nervous system insulin resistance, however, is more difficult to assess, while a clear-cut definition is thus far lacking. Previous studies have demonstrated that whole-body insulin resistance in obese subjects is accompanied with higher brain glucose-uptake (BGU) during the insulin clamp, compared to lean controls, and that BGU increases from the fasting to the insulin clamp state. On the contrary, there is no difference in BGU under fasting conditions between obese subjects and healthy lean controls. No previous studies have evaluated brain glucose uptake in clamp conditions in subjects with MCI or early AD.

The aim of this study is to evaluate if brain glucose uptake is increased in MCI/ early AD subjects in a similar manner as in morbidly obese subjects in an insulin-stimulated state (during a hyperinsulinemic clamp) when compared to the fasting state, and when compared to controls. The investigators hypothesize that MCI subjects would have CNS insulin resistance that could, in time, contribute to the pathological process of AD.

The investigators will recruit altogether 20 MCI subjects from the local memory clinic, and healthy controls through advertisements. All participants will undergo two [18F]-fluorodeoxyglucose (FDG) positron emission tomography (PET) scans (one in the fasting state and one during the hyperinsulinemic clamp), a magnetic resonance image scan for structural changes, blood sampling, and comprehensive cognitive testing. The participants will also undergo a [11C]PIB-PET scan to measure brain amyloid accumulation.

Understanding the metabolic changes in the brain preceding AD could help in developing disease-modifying treatments in the future.

DETAILED DESCRIPTION:
Alzheimer´s disease (AD) and other diseases causing dementia have become increasingly important causes of disability in elderly people worldwide. Mainly due to a rise in life-expectancy, the prevalence of dementia is estimated to double during the next 15 years.

Despite the acknowledgement of the global burden of persons with dementia and intensive research in the field, no curing treatment is yet available for AD or the less common forms of dementia. It seems that insulin resistance would be an important link between diabetes and dementia. Thus, research focusing on the cognitive and the neuropathological changes associated with insulin resistance is needed to evaluate if insulin resistance is an independent risk factor for cognitive decline and dementia, and more specifically, AD. Insulin has many important functions in the central nervous system (CNS). Insulin is actively transported through the blood-brain barrier (BBB) by a transporter in a saturable manner. In addition to transporting insulin from the blood flow to the CNS, the insulin-binding sites act as receptors and activate intra-cellular signaling cascades that alter the functions of the BBB cells in numerous ways.

Insulin resistance has been traditionally thought to occur mainly in the muscles, the liver, and in adipocytes. The brain has been considered an insulin insensitive organ, mainly because glucose uptake in the brain is thought to be mostly independent of insulin. In recent years, however, evidence of insulin resistance occurring also in the CNS has started to accumulate. In obese rodents the binding of insulin to the endothelium of the BBB was reduced when compared to lean animals, and plasma insulin levels correlated negatively to specific insulin binding in the BBB. A similar inverse relationship was found between higher plasma insulin and a lower number of insulin receptors in the liver, suggesting that peripheral hyperinsulinemia downregulates the expression of insulin receptors at the BBB in a similar way as in the peripheral tissues. A magnetoencephalographic study showed that in obese humans the cerebrocortical response to infused insulin during a hyperinsulinemic euglycemic clamp was reduced when compared to lean individuals. These results indicate that peripheral hyperinsulinemia leads to a reduced insulin response in the brain, probably due to lower insulin concentrations in the CNS as a result of insulin transporter down-regulation at the BBB.

In addition to the direct effects of insulin resistance on AD neuropathology, insulin resistance has negative effects on cerebrovascular function. The metabolic syndrome - of which insulin resistance is the key feature - is associated with an increased risk of stroke and brain white matter lesions. The brain is highly dependent of adequate microvascular blood flow, which is maintained by vascular reactivity, and mediated by nitric oxide and endothelial function. Individuals with insulin resistance have been shown to have lower cerebral blood flow in the cortex than normal controls. The vascular injuries associated with insulin resistance might promote the neuropathological changes of AD by, for example, disturbing Aβ transportation between the CNS and periphery. In turn, Aβ deposits in the blood vessel wall can induce inflammation thereby damaging the endothelium. To summarize, insulin resistance is linked to vascular cognitive impairment through brain vascular lesions which, in turn, might be a "second hit" that contributes to the clinical symptoms of AD in the presence of AD neuropathological changes, i.e. Aβ and neurofibrillary tangles.

Measuring brain insulin resistance The definition of systemic insulin resistance is based on tissue-level studies whereseveral molecular defects have been established. For obvious reasons, such studies cannot be performed in the human brain in vivo to define central insulin resistance (IR). To date, there is no consensus on how to measure insulin resistance in the central nervous system in humans. Considering that both systematic and CNS IR have been linked to cognitive decline and AD, many groups have attempted to demonstrate IR in the human brain with different methods.

A seminal post-mortem study demonstrated insulin resistance at tissue level in the brains of patients with AD. They showed that in the neurons of AD brains the response to insulin incubation by the neuronal insulin receptors and the signaling cascades following insulin receptor activation was attenuated when compared to cognitively normal controls and MCI subjects, and that these differences were independent of diagnosis of T2D before death. More recently, a group led by Kapogiannis used neuronally derived extracellular vesicles extracted from plasma to demonstrate defects in insulin signaling in AD patients when compared to controls.

Although brain glucose uptake is thought to be mostly independent of circulating levels, studies performed at the Turku PET Centre have consistently shown that systemic insulin resistance (as demonstrated with the hyperglycemic euglycemic clamp) is associated with elevated brain glucose uptake, measured with [18F]FDGPET during the euglycemic clamp. The investigators therefore propose that elevated brain [18F]-FDG uptake during the euglycemic clamp could be used as a proxy for CNS insulin resistance.

Aims The aim of the present study is to evaluate if i) MCI due to AD is associated with central nervous system insulin resistance, measured with brain [18F]FDG-PET scanning during the euglycemic clamp (compared to a fasting state [18F]FDG-PET scan in the same individuals) ii) MCI due to AD is accompanied by central nervous system insulin resistance, when compared to age- and sex-matched cognitively normal individuals iii) either whole-body insulin resistance or CNS insulin resistance is associated with cognitive performance, measured with comprehensive cognitive tests in a) MCI patients; b) cognitively unimpaired individuals iv) either whole-body insulin resistance or CNS insulin resistance is associated with brain amyloid accumulation, measured with [11C]PIB-PET, or with biomarkers of Alzheimer's disease (phospho-tau 181, phospho-tau 231, total tau, glial fibrillary acidic protein, neurofilament light chain), measured from plasma

Methods Study population and recruitment The investigators will recruit altogether 20 study volunteers with a diagnosis of MCI due to AD or early AD or episodic memory decline during the last 6 months from the local memory clinics and by contacting doctors who treat and diagnose memory disorders. Recruitment will also be performed via advertisements.

Study protocol The participants will be examined at the Turku PET Centre. The study will require approximately 4 study visits.

Study visit 1 (screening and oral glucose tolerance test) The participants will be asked to arrive at the Turku PET Centre after an overnight fast (minimum 10 hours). The study volunteers will be asked to sign the written consent forms containing information on the study procedures. The forms will be sent to the participants before the first study visit by mail or email. After signing the informed consent the participants will be thoroughly interviewed (medical history, medication, smoking, alcohol usage, educational history, depressive symptoms). Weight, height and blood pressure will be measured, and the participants will undergo a neurological and a physical examination. The participants' family member or a close friend will be asked to accompany the participant on the first visit, and to fill in the clinical rating scale (CDR) forms. A standard 75-g oral glucose tolerance (OGTT) will be performed with frequent sampling (every 30 minutes) for plasma glucose, insulin and C-peptide.

Study visit 2 cognitive testing and [11C]PIB-PET scan A neuropsychological investigation assessing memory and other cognitive domains will be performed by a trained psychology student. The duration of the testing is approximately 1,5 hours. In addition, all participants will undergo computerized cognitive testing which lasts approximately for 1 hour. If in the testing clinically significant abnormalities are seen the study participants will be directed to further investigations via regular health care system.

All participants will undergo a [11C]PIB-PET scan of the brain, to estimate brain beta-amyloid accumulation, one of the earliest signs of AD. 500 MBq of [11C]PIB will be injected intravenously, after which the participants are instructed to lie down for 30 minutes. After 40 minutes the participants are positioned inside the PET camera. The scan duration is 50 minutes (40 to 90 minutes).

Study visit 3 (fasting [18F]-FDG PET scan and MRI scan) The participants will be asked to arrive at the Turku PET Centre after an overnight fast (minimum 10 hours).

Structural brain and whole body MRI will be performed to obtain anatomical reference. The investigators will use the MR part of a 3T PET-MR system for the study (Philips Ingenuity TF, Philips Healthcare, OH, USA).

After the completion of the brain MRI/MRS studies, an intravenous line will be inserted. Fasting plasma glucose will be measured (because hyperglycemia fP-gluk > 9 mmol/l may affect FDG-PET scanning) and fasting venous blood samples will be drawn. The participants will then receive an intravenous injection of 100 MBq [18F]-FDG. After the injection they will undergo dynamic PET imaging (scan duration 60 minutes) as described in detail below.

Study visit 4 (hyperinsulinemic euglycemic clamp [18F]-FDG PET scan) Hyperinsulinemic, euglycemic clamp technique will be used to promote tissue glucose uptake and measure insulin sensitivity. Initially, two cannulas will be inserted, one in a radial or an antecubital vein for PET tracer injection and infusion of glucose and insulin, another in the opposite radial or antecubital vein for blood sampling. In the clamp study subjects are administered intravenous insulin at a steady rate of 40 mU/m2/min and normoglycemia is maintained using a variable rate infusion of 20 % glucose based on plasma glucose measurements, which are performed every 5-10 min from arterialized venous blood. The investigators will also collect samples to determine plasma insulin, serum free fatty acid and metabolic biomarkers during the study.

The clamp will be performed together with [18F]-FDG-PET/CT. Whole-body glucose uptake (M-value) is presented as the average of three to four 20-minute periods during steady euglycemia. An urine sample will be collected after the scanning to measure tracer lost in urine for the calculation of endogenous glucose production.

Whole-body scan with [18F]-FDG and PET/CT After 60 minutes from the start of clamp and when steady euglycemia (plasma glucose 5.0 ± 0.5 mmol/L) is reached, the subjects will be injected intravenously with 100 MBq of [18F]-fluorodeoxyglucose ([18F]-FDG). Thereafter [18F]-fluorodeoxyglucose uptake in the brain and whole body will be measured using a combined clinical total body PET/CT camera (Quadra). To obtain arterial input, samples or plasma radioactivity will be collected through the study and measured with an automatic gamma counter (Wizard 1480 3", Wallac, Turku, Finland). The scan will last for 60 minutes. Tissue activity and fractional uptake will be calculated by using graphical analysis.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for MCI/early AD -patients for the present study are:

* diagnosis of MCI due to AD or early AD based on a neurologist's or a geriatrician's clinical examination and/ or cognitive testing showing either a decline during at least a 6 month follow-up or a slight decline in episodic memory
* clinical dementia rating (CDR) = 0,5, based on an interview with the patient's spouse or close relative
* age 55 to 80 years
* Inclusion criteria for the cognitively unimpaired group for the present study are:
* no subjective cognitive complaints
* consortium to establish a registry for Alzheimer´s Disease (CERAD) test battery at screening visit within the normal range
* clinical dementia rating (CDR) = 0, based on an interview with the study volunteer´s spouse or close relative
* age 55 to 80 years

Exclusion Criteria:

Exclusion criteria for both groups are:

* diabetes (type 1 or type 2)
* overweight or obesity (BMI > 26 kg/m2)
* BMI < 18 kg/m2
* impaired fasting glucose of impaired glucose tolerance in the 2-hour oral glucose tolerance test, performed at the screening visit
* other major neurological disease than MCI (such as a major stroke, multiple sclerosis, Parkinson's disease). Volunteers with minor neurological diseases such as migraine and a previous transient ischemic attack (TIA) can participate
* major psychiatric illness such as schitzophrenia, bipolar disorder or major depression
* conditions that affect the ability to participate in PET or MRI scanning (cancer diagnosis/ treatment within the last five years, claustrophobia, metal object in the body)

Exclusion criteria for the MCI/early AD patients only are:

• amyloid negative PET scan (during the study or performed previously in the clinic or normal beta-amyloid42 or beta-amyloid42/40 ratio in CSF (measured previously in the clinic) (to exclude patients with cognitive decline due to some other pathological process than AD)

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit 20 volunteers with a diagnosis of MCI due to AD or early AD or episodic memory decline during the last 6 months from the local memory clinics and by contacting doctors who treat and diagnose memory disorders. Recruitment will also be performed via. Inclusion will be made at the first screening visit. Patients with Alzheimer´s dementia - i.e. cognitive impairment severe enough to cause problems in activities of daily living - will not be included in the study due to the study protocol which requires co-operation and the ability to lie still in the PET scanner for approximately 60 minutes.
  The investigators will also recruit 20 cognitively unimpaired controls.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Brain glucose uptake | 0 months
  Differences in brain glucose uptake (umol/100ml/min) measured during insulin clamp conditions between the two groups.

SECONDARY OUTCOMES:
[11C]PIB-PET brain uptake | 0 months
  Differences in [11C]PIB-PET brain uptake (in standardized uptake value) between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Ekblad, MD, Principal Investigator — Turku PET Centre
Locations (1):
- Turku PET Centre, Turku, Finland

IPD SHARING:
Plan to Share IPD: No
Some datasets generated during and/or analyzed during the current study may not be publicly available but are available from the corresponding author on reasonable request.